CLINICAL TRIAL: NCT01482260
Title: Comparative Microarray Analysis of microRNA Expression Profiles in Primary Cutaneous Malignant Melanoma, Cutaneous Malignant Melanoma Metastases and Benign Melanocytic Naevi
Brief Title: Comparative Microarray Analysis in Primary Cutaneous Malignant Melanoma
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Michael Sand, Principal Investigator, Ruhr University of Bochum
Other Study IDs: microRNA5
Record Dates: First submitted 2011-11-26; First posted 2011-11-30 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Cutaneous Malignant Melanoma
MeSH Terms: conditions — Melanoma, Cutaneous Malignant | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — skin biopsy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Primary Cutaneous Malignant Melanoma
  Interventions: Procedure: Biopsy
- Cutaneous Malignant Melanoma Metastases
  Interventions: Procedure: Biopsy
- Benign Melanocytic Nevi
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Biopsy

SUMMARY:
Perturbations in microRNA (miRNA) expression profiles has been reported for cutaneous malignant melanoma (CMM). This study will be an exploratory analysis by miRNA expression profiling using microarrays.

DETAILED DESCRIPTION:
Perturbations in microRNA (miRNA) expression profiles has been reported for cutaneous malignant melanoma (CMM). With regards to a rapidly growing number of newly discovered miRNA sequences, the availability of up-to-date miRNA expression profiles for primary cutaneous malignant melanoma (PCMM), cutaneous malignant melanoma metastases (CMMM) and benign melanocytic naevi (BMN) is limited. Patients with PCMM, CMMM and BMN are included in the study to perform an exploratory analysis by miRNA expression profiling using microarrays. Expression levels of miRNA candidates will be validated by TaqMan real-time quantitative polymerase chain reaction (RT-PCR).

ELIGIBILITY:
Inclusion Criteria:

* Primary Cutaneous Malignant Melanoma
* Cutaneous Malignant Melanoma Metastases
* Benign Melanocytic Naevi

Exclusion Criteria:

- Other Skin Cancer than Primary Cutaneous Malignant Melanoma

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with
  * Primary Cutaneous Malignant Melanoma
  * Cutaneous Malignant Melanoma Metastases
  * Benign Melanocytic Naevi
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-12; Primary Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Falk G Bechara, PD Dr., Study Director — Department of Dermatology, Venereology and Allergology, Ruhr-University Bochum; Peter Altmeyer, Prof. Dr., Study Chair — Department of Dermatology, Venereology and Allergology, Ruhr-University Bochum
Locations (1):
- Department of Dermatology, Venereology and Allergology, Ruhr-University Bochum, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Sand M, Skrygan M, Sand D, Georgas D, Gambichler T, Hahn SA, Altmeyer P, Bechara FG. Comparative microarray analysis of microRNA expression profiles in primary cutaneous malignant melanoma, cutaneous malignant melanoma metastases, and benign melanocytic nevi. Cell Tissue Res. 2013 Jan;351(1):85-98. doi: 10.1007/s00441-012-1514-5. Epub 2012 Oct 31. PMID 23111773